CLINICAL TRIAL: NCT02982642
Title: The Safety and Efficacy of 1612 Capsules in Treatment of aMnestic Mild Cognitive Impairment: a 52-week, Double Blind,Randomized, Parallel,Placebo Controlled Trial.
Brief Title: Efficacy and Safety of 1612 Capsules in aMnestic Mild Cognitive Impairment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor cannot conduct research due to insufficient funding supportment
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Clinical Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z20055424
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1612 capsule (Experimental): Subjects will take 1612 capsule 3 capsules per time(0.38g per capsule), 3 times per day for 52 weeks
  Interventions: Drug: 1612 capsule
- Placebos (Placebo Comparator): Subjects will take palcebo identified to 1612 capsule 3 capsules per time, 3 times per day for 52 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 1612 capsule — Subjects will be assigned 1612 capsule,3 capsules per time(0.38g per capsule), 3 times per day.1612 capsule is a Chinse herbal medicine,which can tonification of spleen and kidney, mainly contains shudihuang(Rehmannia glutinosa),shanyao(Dioscorea opposita),shichangpu(Uncaria rhynchophylla)and so on,
  Arms: 1612 capsule
Drug: Placebos — Subjects will be assigned placebo identified to 1612 capsule,3 capsules per time, 3 times per day
  Arms: Placebos

SUMMARY:
This study is a 52-weeks, multicenter, randomized, double-blind, placebo controlled, parallel trial which will be carried out in 15 centers around China. The study population includes amnestic mild cognitive impairment patients (planned a total of 240) aged 55-85 in both gender. Participants will be randomly allocated to 1612 capsules (1.14g per time, 3 times per day) or placebo for a 52-weeks double-blind treatment period. The primary outcome measure is change from baseline in the Alzheimer's Disease Assessment Scale- Cognition Subscale (ADAS-cog) and rate of conversion to dementia. The secondary outcomes are changes from baseline in the Mini-Mental State Examination (MMSE), Delayed Story Recall test (DSR), Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24). Safety is being assessed by observing side effects and adverse reaction during the entire treatment period. Statistical analysis will be conducted according to per-protocol population and intend-to-treat population and the safety will be analyzed in safety set.

ELIGIBILITY:
Inclusion Criteria:

Patients should be enrolled if they met the following criteria[14]:

1. cognitive complaints from the patients or their families;
2. objective evidence for memory impairment, delayed story recall test(DSR)<12.6(age50-64 less than15.5,65-74less than 12.5,older 75 less than10);
3. normal general cognitive function, with Mini-Mental State Examination (MMSE) score of between 24 and 30 (including 30);
4. preservation of activities of daily living, with Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24) score between 38 and 52;
5. cognitive disorders as evidenced by clinical evaluation, with clinical dementia rating scale=0.5,memory domain = 0.5;
6. absence of dementia, not sufficiently impaired cognitively and functionally to meet DSM-IV criteria,
7. enough vision and hearing to accomplishment neuropsychological test;
8. capability to read words and write simple sentence;
9. capability and willingness to give informed consent and to comply with the study procedures.

Exclusion Criteria:

The patients would be ineligible if they had the following conditions:

1. non amnestic Mild cognitive impairment;
2. meeting the diagnostic criteria for dementia;
3. cognitive impairment resulting from conditions such as acute cerebral trauma, cerebral damage due to a lack of oxygen, epilepsy vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor ,or drug abuse or alcohol abuse
4. having significant psychiatric disease, depression, the Hamilton depression scale >12; CT or MRI scan showed central nervous system infections Infarction or focal lesions within 12 months，the Hachinski Ischemic Scale (HIS)>4;
5. combined following disease: diabetes; poor controlled hypertension or severe arrhythmias; or suffered from heart infarction within 3 months; severe asthma or COPD; severe indigestion; gastrointestinal tract obstruction; gastroduodenal ulcer;
6. used cholinesterase inhibitors or memantine within 1 month;
7. history of hypersensitivity to the treatment drugs;
8. concomitant drugs with the potential to interfere with cognition;
9. administration of other investigational drugs; severe impairment of the functions of the kidney or liver;
10. vegetarians or contraindications for animal innards.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive scores: Alzheimer Disease Assessment Scale-cognitive subscale (ADAS-cog) | 52 weeks
  Cognition will accessed with the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog), at baseline (day 1 clinic visit) and week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of rate of dementia conversion from mild cognitive impairment | 52 weeks
  The rate of demention conversion will accessed from baselin at week 0 and week 4, week 12, week 24 ,week 36 , week 48 and week 52.

SECONDARY OUTCOMES:
Change from baseline to end of double-blind treatment of Mini-Mental State Examination(MMSE) | 52 weeks
  Cognition will accessed with the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog), at baseline (day 1 clinic visit) and week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of Delayed Story Recall test (DSR) | 52 weeks
  Memory will accessed with the delayed story recall test(DSR), at baseline (day 1 clinic visit) and week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24) | 52 weeks
  Ability of daily living will accessed with the Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24), at baseline (day 1 clinic visit) and week 4, week 12, week 24 ,week 36 , week 48 and week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, M.D,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No